CLINICAL TRIAL: NCT03778606
Title: Oligosaccharide Supplementation Among Hematology-Oncology Clostridium Difficile Colonized Patients
Brief Title: Oligosaccharide for Cdiff(+) Heme-onc Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Silvia Munoz-Price, Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO00033794
Record Dates: First submitted 2018-11-30; First posted 2018-12-19 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Clostridium Difficile; Hematologic Diseases
Keywords: Clostridium difficile; Asymptomatic carrier; Potato starch; Non digestable oligosaccharide
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Potato starch supplementation (Experimental): Twelve patients found to be colonized with C. difficile will undergo twice a day potato starch supplementation.
  Interventions: Dietary Supplement: Potato starch

INTERVENTIONS:
Dietary Supplement: Potato starch — Potato starch will be given twice a day for up to 14 days, discharge, or death, whichever occurs first.

SUMMARY:
Clostridium difficile causes ~453,000 infections and ~29,300 deaths per year in the US, making it the most common hospital acquired infection in the country. C. difficile is an anaerobic bacterium that has the capacity to inhabit the colon of humans and other mammals. Initially thought to be a commensal, it was later found to be associated with antibiotic induced enterocolitis. Since then, it has gradually become one of the most important healthcare associated pathogens. C. difficile infection (CDI) causes colitis, which is inflammation of the colonic mucosa with a spectrum of severity from mild to more protracted diarrhea, abdominal pain, fever, toxic megacolon, sepsis, and in some instances death. Mortality occurs despite the existence of three antibiotic options. CDI is also associated with higher hospital readmission rates, and associated healthcare costs in the US are estimated at 4.8 billion dollars annually. Due to the significance of C. difficile in healthcare, hospital level C. difficile rates are publically reported and closely scrutinized by the Centers for Medicare and Medicaid. Standard infection control bundles are proving to be insufficient for controlling the national C. difficile problem. Better understanding of the biological steps preceding clinical infection and reversal of the underlying gut dysbiosis will allow us to curtail our C. difficile epidemic. The present study aims to manipulate the gut microbiota to halt the biological progression of C. difficile.

CDI is a serious problem in hematology-oncology patients. The incidence of CDI in the hematology-oncology population is much higher than in other populations and hematology-oncology inpatient units frequently have the highest incidence of CDI cases within an institution. Additionally, hematology-oncology patients have high rates of C. difficile colonization upon hospitalization and more than 50% of patients detected with C. difficile colonization before bone marrow transplantation end up diagnosed with hospital associated CDI. This finding is not trivial as CDI treatment with oral vancomycin causes major and prolonged perturbations of their intestinal microbiota, which has been associated with higher mortality. In addition to the usual complications of CDI, a higher incidence of graft-versus-host-disease has been described in patients with CDI.

DETAILED DESCRIPTION:
Aim 1/Objective 1. Establish the feasibility of oligosaccharide supplementation and twice a week stool collections among 12 C. difficile colonized hematology-oncology inpatients. It will be determined if at least 70% of the oligosaccharide dosages are taken by at least 8 (>=66%) of the 12 enrolled patients. Additionally, the ability to collect at least 50% of the scheduled stool samples will be evaluated.

Aim 1 will provide important information about the ideal food/drink to mix the potato starch supplemented in this study. The knowledge gained in this pilot will be used to design a future phase II or III clinical trial.

Aim 2. Explore the impact of oligosaccharide supplementation on C. difficile loads and relative abundance of Firmicutes. All stool samples will undergo 16S ribosomal ribonucleic acid (rRNA) and bioinformatics at the MCW's Genomic and Precision Medicine Center and C. difficile quantitative polymerase chain reaction (qPCR) at the PI's research laboratory. Historical controls will be obtained from a group of over 450 hematology-oncology inpatients who underwent at least one C. difficile surveillance test and whose stool samples are currently being processed for 16S rRNA by the PI's team. Controls at a 3:1 ratio with cases will be matched based on underlying disease, unit of admission, antibiotic use, baseline C. difficile fecal loads, and baseline relative abundance of Firmicutes.

Objective 2a. Evaluate the impact of oligosaccharide supplementation on the change of C. difficile fecal loads when compared to historical controls.

Objective 2b. Explore the effect of oligosaccharide supplementation on the change in relative abundance of Firmicutes when compared to historical controls.

It is expected a reduction will occur in C. difficile fecal loads during oligosaccharide supplementation when compared to matched controls. Conversely, it is expected an increase in the relative abundance of Firmicutes (or some of its operational taxonomic units; OTUs) during oligosaccharide replacement will occur when compared to matched controls. The knowledge gained with Objectives 2a and 2b will be used to determine the sample size needed to design future phase II or phase III clinical trials.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all inclusion criteria to be eligible to participate in the study.

* Patients must be at least 18 years of age at time of consent.
* Positive C. difficile surveillance test.
* Absence of diarrhea or abdominal pain within the past 48 hours.
* Patient admitted in a hematology-oncology unit which for the purposes of this study will be defined as 7-CFAC and 8-CFAC.

Exclusion Criteria:

Patients must NOT meet any exclusion criteria to be eligible to participate in the study.

* Presence of >= grade I nausea/vomiting.
* Inability to take oral medications or food.
* Expected length of hospitalization or survival less than 5 days
* Patient is only boarding in hematology-oncology units and would have not otherwise been admitted to these units.
* Unwillingness or inability to provide written informed consent.
* Women known to be pregnant or lactating during the study.
* History of inflammatory bowel disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Stool samples will be collected twice a week while on potato starch supplementation and 1 time at 7-days post- starch supplementation to assess any changes in the frequency of collection during the 21-day period. | Day 1- Day 21
  Samples will be collected twice a week (4-5 times during supplementation) and one time at day 21 or discharge, whichever happens first.
Oligosaccharide intake assessed by a patient diary to measure supplementation feasibility | Day 1-Day 14
  Patients will be provided with a diary in which they will document compliance with oligosaccharide intake. It is anticipated ≥70% of intended doses to be fully administered by the patient.
The feasibility of collecting all available stool samples stool will be assessed. A rate ≥50% of correctly collected and processed samples will be considered feasible. | Day 1-Day 14
  It is expected ≥50% of stool samples to be correctly collected and processed.

SECONDARY OUTCOMES:
Changes in C. difficile loads will be assessed using C. difficile quantitative polymerase chain reaction (qPCR). | Day 1-Day 14
  Stool samples collected for diagnosis and any additional stool collections will be thawed in batches and one cc aliquot will be extracted refreezing the remaining sample at -80 degrees F. One cc aliquot will then be divided into 4 sub-samples of equal volume and with the same unique identifier. This identifier will be able to chronologically cluster samples by each unique patient. A sample will be used for C. difficile qPCR quantitative determination.
Changes in Firmicutes' relative abundance due to oligosaccharide supplementation measured by 16S rRNA gene sequencing | Day 1-Day 14
  Sub-sample of stool from diagnosis, and additional stool collections will be used for 16S ribosomal ribonucleic acid gene sequencing to determine the microbiome community structure

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided